CLINICAL TRIAL: NCT03309904
Title: Sport Without Injury ProgrammE Floorball
Acronym: SWIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Martin Hägglund, Associate professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHägglund SWIPE Floorball
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Parallell group cluster-randomized trial
Who Masked: Outcomes Assessor
Masking Description: Statistician performing outcome analyses are blinded to group belonging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee Control training program (Experimental): The Knee Control program is a neuromuscular training program that consists of 6 different exercises, with 4 levels of progression and one pair-exercise, for each exercise. The Knee Control program takes about 10 minute to complete after familiarization. In addition, a 5-minute running warm-up is instructed to coaches. Coaches are to perform the Knee Control program + the 5 minute warm-up at all training sessions during the season, and the 5 minute warm-up before all matches.
  Interventions: Other: Knee Control training program
- Control group - usual training (No Intervention): The control group teams receive no intervention, and coaches are instructed to carry out their normal training and warm-up practice throughout the season.

INTERVENTIONS:
Other: Knee Control training program — 10-minute training program to be performed at all team training sessions during the season.
  Arms: Knee Control training program

SUMMARY:
This study evaluates the preventive effect of a neuromuscular training program on injuries in youth floorball players. Half of participants will receive the training program, and half act as control and perform their usual training practices.

DETAILED DESCRIPTION:
The study is a cluster-randomized controlled trial including male and female youth (12-17 years) floorball players. Club is used as cluster unit.

Coaches in the intervention group receive education of the preventive neuromuscular training program Knee Control (Knäkontroll) before the start of the season. Knee Control consists of 6 different exercises, with 4 different variations and 1 pair-exercise, and takes about 10 minutes to complete. In addition, coaches are instructed to perform a 5-minute running warm-up before the Knee Control exercises. Teams are to carry out the intervention at all training sessions, and the 5-minute warm-up also before all matches.

Coaches in the control group carry on their normal training and warm-up routines with their clubs.

Teams are followed for one full season: October 2017 - March 2018. Data registered for the study include exposure to floorball training and matches, and injuries that occur as a result of participation in floorball.

ELIGIBILITY:
Inclusion Criteria:

* Teams with players 12-17 years of age (born 2000-2005)
* Teams who have not used a structured training program aiming to prevent injuries (the Knee Control or similar program) on a regular basis the last year
* Teams who have training at least twice per week

Exclusion Criteria:

-

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 910 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
All physical complaints injury | Study start up to end of season (6 months)
  Any floorball related injury regardless of need of care or absence from floorball training or matches ("all physical complaints" injury definition)

SECONDARY OUTCOMES:
Time-loss injury | Study start up to end of season (6 months)
  Floorball related injury causing absence from the next training or match with the team ("time-loss injury")
Medical attention injury | Study start up to end of season (6 months)
  Floorball related injury requiring the player to seek care ("medical attention injury")
Adverse events | Study start up to end of season (6 months)
  Adverse events of using the program (intervention group only)
Intervention compliance and fidelity | Study start up to end of season (6 months)
  Coach reported compliance and fidelity with the program protocol (intervention group only)
Coach experience of injuries and intervention program | Baseline and 6 months
  Coach baseline and follow-up experiences of injuries (control group and intervention group) and of the Knee Control program (intervention group only)
Player experience of injuries and intervention program | Baseline and 6 months
  Player baseline and follow-up experiences of injuries (control group and intervention group) and of the Knee Control program (intervention group only)
Exercise fidelity | At approximately 2 months and 5 months
  Exercise fidelity (observation of the technique when using the intervention in select intervention group teams)
Health care need | After study end at 6 months
  Number of health care visits due to floorball related injuries during the season, type of diagnostic examinations and treatments
Costs | After study end at 6 months
  Estimated costs of floorball related injuries and costs of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hägglund, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Undecided, possibly share deidentified exposure and injury outcome data

REFERENCES:
- [Derived] Sonesson S, Dahlstrom O, Panagodage Perera NK, Hagglund M. Risk factors for injury and illness in youth floorball players - A prospective cohort study. Phys Ther Sport. 2023 Jan;59:92-102. doi: 10.1016/j.ptsp.2022.11.008. Epub 2022 Dec 5. PMID 36528005
- [Derived] Perera NKP, Walden M, Lindblom H, Akerlund I, Sonesson S, Hagglund M. Illness prevalence and symptoms in youth floorball players: a one-season prospective cohort study involving 471 players. BMJ Open. 2021 Dec 14;11(12):e051902. doi: 10.1136/bmjopen-2021-051902. PMID 34907058
- [Derived] Akerlund I, Walden M, Sonesson S, Hagglund M. Forty-five per cent lower acute injury incidence but no effect on overuse injury prevalence in youth floorball players (aged 12-17 years) who used an injury prevention exercise programme: two-armed parallel-group cluster randomised controlled trial. Br J Sports Med. 2020 Sep;54(17):1028-1035. doi: 10.1136/bjsports-2019-101295. Epub 2020 Jan 28. PMID 31992545